CLINICAL TRIAL: NCT07190430
Title: A Phase 1, Open-label, Fixed Sequence Study to Evaluate The Effect of Steady-State Dosing of PF-08049820 on the Single Dose Pharmacokinetics of Oral Contraceptives, Midazolam, and Dabigatran in Healthy Adult Female Participants
Brief Title: A Study to Learn If the Study Medicine Called PF-08049820 Changes How the Body Processes the Other Study Medicines Called Oral Contraceptives, Midazolam, and Dabigatran in Healthy Adult Female Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C6231004
Record Dates: First submitted 2025-09-02; First posted 2025-09-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Healthy Volunteers
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Midazolam; Dabigatran; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Baseline Midazolam (Other): Participants will receive a single dose of 2 mg midazolam in the morning on Day 1
  Interventions: Drug: Midazolam
- Baseline dabigatran etexilate (Other): Participants will receive a single dose of 150 mg dabigatran etexilate in the morning on Day 1
  Interventions: Drug: Dabigatran Etexilate
- Baseline oral contraceptives (Other): Participants will receive a single dose of Portia (30 mcg of ethinyl estradiol (EE) and 150 mcg of levonorgestrel (LN)) or equivalent oral tablet in the morning on Day 1
  Interventions: Drug: Portia (EE and LN) or equivalent oral tablet
- Drug Drug Interaction (DDI) midazolam (Experimental): Participants will receive a single dose of 2 mg midazolam in the morning on Days 2 and 10 only with PF-08049820 Days 1 to 10
  Interventions: Drug: PF-08049820; Drug: Midazolam
- DDI dabigatran etexilate (Experimental): Participants will receive a single dose of 150 mg dabigatran etexilate in the morning on Day 1 only with PF-08049820 Days 1 to 2
  Interventions: Drug: PF-08049820; Drug: Dabigatran Etexilate
- DDI oral contraceptives (Experimental): Participants will receive a single dose of Portia (30 mcg of EE and 150 mcg of LN) or equivalent oral tablet in the morning on Day 1 only with PF-08049820 on Days 1 to 2
  Interventions: Drug: PF-08049820; Drug: Portia (EE and LN) or equivalent oral tablet

INTERVENTIONS:
Drug: PF-08049820 — Administered orally
  Arms: DDI dabigatran etexilate; DDI oral contraceptives; Drug Drug Interaction (DDI) midazolam
Drug: Midazolam — Administered orally
  Arms: Baseline Midazolam; Drug Drug Interaction (DDI) midazolam
Drug: Dabigatran Etexilate — Administered orally
  Arms: Baseline dabigatran etexilate; DDI dabigatran etexilate
Drug: Portia (EE and LN) or equivalent oral tablet — Administered orally
  Arms: Baseline oral contraceptives; DDI oral contraceptives

SUMMARY:
The purpose of this study is to see how a medicine called PF-08049820 affects how other medicines move through the body. This information will help plan future studies. The other medicines include:

* Birth control pills (containing ethinyl estradiol and levonorgestrel)
* Midazolam (used to help people relax or sleep)
* Dabigatran etexilate (used to prevent blood clots)

This study is seeking participants who:

* are female and are 18 years or older
* weigh more than 110 pounds (50 kg)
* have a healthy body weight (not too low or too high)
* are generally healthy with no serious medical problems. People with serious health problems, recent medicine use, or who had certain vaccines recently cannot join.
* are willing to follow all the study rules The study has 6 parts, and each part happens one after the other. In the first 3 parts, participants take just one dose of each medicine (midazolam, dabigatran, and birth control pills) to see how these medicines work alone. In the last 3 parts, they take PF-08049820 twice a day, along with one of the other medicines, to see how PF-08049820 changes the way those medicines move through the body. The whole study will take about 12 to13 weeks and participants will stay overnight in the clinic for about 25 days.

ELIGIBILITY:
Inclusion Criteria:

* Female participants ≥18 years of age, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* BMI of 16 to 32 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, Hepatitis B surface antigen (HBsAg), Antibody to hepatitis B surface antigen (HBsAb), Hepatitis B core antibody (HBcAb), or Hepatitis C Virus Antibody (HCVAb). A positive HBsAb result and a history of Hepatitis B vaccination is allowed.
* History of thromboembolic diseases.
* History of bleeding tendencies.
* History of myocardial infarction, unstable angina, arterial revascularization, mechanical prosthetic heart valve, stroke, New York Association Functional Class II-IV heart failure, or transient ischemic attack.
* Any known allergy or intolerance to midazolam or other drugs in the benzodiazepine class, and/or to dabigatran etexilate, and/or to OCs.
* Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of certain prescription or nonprescription drugs and dietary (e.g. grapefruit) and herbal supplements within up to 14 days or 5 half-lives, whichever is longer, prior to the first dose of study intervention.
* Recent exposure to live or attenuated vaccines within 28 days of the screening visit.
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of screening.
* Use of tobacco/nicotine containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants ≥18 years of age
Enrollment: 16 (Actual)
Dates: Start 2025-10-03 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the curve (AUC) of Midazolam | From pre-dose up to 24 hours post dose in Periods 1 and 4
PK: Plasma Maximum Concentration (Cmax) of Midazolam | From pre-dose up to 24 hours post dose in Periods 1 and 4
PK: Area Under the curve (AUC) of dabigatran | From pre-dose up to 48 hours post dose in Periods 2 and 5
PK: Cmax of dabigatran | From pre-dose up to 48 hours post dose in Periods 2 and 5
PK: AUC of Ethinyl estradiol and levonorgestrel | From pre-dose up to 96 hours post dose in Periods 3 and 6
PK: Cmax of Ethinyl estradiol and levonorgestrel | From pre-dose up to 96 hours post dose in Periods 3 and 6

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose of study intervention until Follow Up Visit (28 to 35 days after the last dose)
Number of Participants With Clinically Significant Change from Baseline in Laboratory Abnormalities | Baseline to Study Day 24
Number of Participants With Clinically Significant Change from Baseline in Vital Signs | Baseline to Study Day 24
Number of Participants With Clinically Significant Change from Baseline in 12-lead Electrocardiogram (ECG) Findings | Baseline to Study Day 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6231004